CLINICAL TRIAL: NCT01844960
Title: A Prospective Double Blinded Randomised Control Trial Comparing Laparoscopic Single Incision Versus Multiple Incision Adjustable Gastric Band Surgery in Patients With Morbid Obesity
Brief Title: Laparoscopic Single Incision -Vs- Multiple Incision Gastric Band Surgery
Acronym: SIMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/LO/1592
Record Dates: First submitted 2012-08-06; First posted 2013-05-03 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2013-04

CONDITIONS: Surgery; Post-operative Pain; Post-operative Recovery
Keywords: Single Incision Surgery; SILS; Laparoscopic Gastric Band; Morbid Obesity; Bariatric Surgery
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple Incision Gastric Band Insertion (Active Comparator): Current standard surgical approach for laparoscopic gastric band insertion
  Interventions: Procedure: Multiple Incision Gastric Band Insertion
- Single Incision Gastric Band Insertion (Experimental): New surgical approach for gastric band insertion
  Interventions: Procedure: Single Incision Gastric Band Insertion

INTERVENTIONS:
Procedure: Single Incision Gastric Band Insertion — Insertion of gastric band though single abdominal incision
  Arms: Single Incision Gastric Band Insertion
Procedure: Multiple Incision Gastric Band Insertion — Insertion of gastric band though multiple abdominal incisions
  Arms: Multiple Incision Gastric Band Insertion

SUMMARY:
A double blinded randomised control trial comparing the differences between laparoscopic single incision versus multiple port bariatric surgery in morbidly obese patients (BMI>35). Single incision surgery is a new minimally invasive surgical technique requiring the surgeon to operate through one small single incision and is virtually scarless. The traditional laparoscopic approach to abdominal surgery is through multiple small incisions (4-7 ports) across the whole abdomen. This study seeks to identify the risks, benefits and costs of the adjustable gastric band insertion via single incision and multiple incision within the morbidly obese patient group.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients, BMI ≥35 kg/m2
* Undergoing gastric band surgery
* Undergone a pre-weight loss surgery risk assessment
* Fit for anaesthesia and surgery
* Fulfil day surgery criteria
* Full understanding of bariatric procedure, with informed consent of the risks and benefits of laparoscopic single incision and multiple incision surgery

Exclusion Criteria:

* Pregnancy
* History of portal hypertension
* Previous gastric surgery or large hiatus hernia
* Previous laparotomy or bariatric surgery
* Weight >150kg (day surgery limit)
* Unwilling to consider surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pain | first 10 days post-operatively

SECONDARY OUTCOMES:
Time to Discharge | Post-operative ward stay (estimated 2-8 hours)

OTHER OUTCOMES:
Conversion to laparoscopic or open surgery | Intra-operatively
Intraoperative and post-operative complications | During surgery (intraoperative) and first 30 days (post-operative)
Operative time | Skin incision to skin closure (estimated 45 -75 minutes)
Cosmesis | 6 weeks to 6 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Ameet G Patel, MS FRCS, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, Greater London, United Kingdom

REFERENCES:
- [Background] Patel AG, Murgatroyd B, Carswell K, Belgaumkar A. Fundus-first transumbilical single-incision laparoscopic cholecystectomy with a cholangiogram: a feasibility study. Surg Endosc. 2011 Mar;25(3):954-7. doi: 10.1007/s00464-010-1240-6. Epub 2010 Aug 19. PMID 20721587
- [Background] Patel AG, Belgaumkar AP, James J, Singh UP, Carswell KA, Murgatroyd B. Video. Single-incision laparoscopic left lateral segmentectomy of colorectal liver metastasis. Surg Endosc. 2011 Feb;25(2):649-50. doi: 10.1007/s00464-010-1237-1. Epub 2010 Jul 22. PMID 20652322
- [Background] Teixeira J, McGill K, Binenbaum S, Forrester G. Laparoscopic single-site surgery for placement of an adjustable gastric band: initial experience. Surg Endosc. 2009 Jun;23(6):1409-14. doi: 10.1007/s00464-009-0411-9. Epub 2009 Mar 14. PMID 19288157
- [Background] de la Torre RA, Satgunam S, Morales MP, Dwyer CL, Scott JS. Transumbilical single-port laparoscopic adjustable gastric band placement with liver suture retractor. Obes Surg. 2009 Dec;19(12):1707-10. doi: 10.1007/s11695-009-9896-5. PMID 19579051
- [Background] Nguyen NT, Slone J, Reavis K. Comparison study of conventional laparoscopic gastric banding versus laparoendoscopic single site gastric banding. Surg Obes Relat Dis. 2010 Sep-Oct;6(5):503-7. doi: 10.1016/j.soard.2009.10.001. Epub 2009 Nov 10. PMID 19969508
- [Background] Tsimoyiannis EC, Tsimogiannis KE, Pappas-Gogos G, Farantos C, Benetatos N, Mavridou P, Manataki A. Different pain scores in single transumbilical incision laparoscopic cholecystectomy versus classic laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2010 Aug;24(8):1842-8. doi: 10.1007/s00464-010-0887-3. Epub 2010 Feb 20. PMID 20174950
- [Background] Patel AG, Murgatroyd B, Ashton WD. Single incision laparoscopic adjustable gastric banding: 111 cases. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):747-51. doi: 10.1016/j.soard.2011.06.013. Epub 2011 Jul 13. PMID 21890429